CLINICAL TRIAL: NCT05265156
Title: An Evaluation of the Tolerability and Acceptability of a New Plant-based Formula for Young Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: High drop out rate
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SBB20R&31559
Record Dates: First submitted 2021-12-16; First posted 2022-03-03 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Healthy Young Children

STUDY DESIGN:
Intervention Model Description: Single arm, prospective, open-label, longitudinal, interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plant based formula for young children (Other): The study is designed with a single arm, so all subjects will receive the study product.
  Interventions: Other: Plant based formula for children aged between 12 and 36 months

INTERVENTIONS:
Other: Plant based formula for children aged between 12 and 36 months — Daily intake of plant based formula for 3 weeks (400ml-600ml per day).

SUMMARY:
An evaluation of the tolerability and acceptability of a new plant-based formula in 45 healthy young children

DETAILED DESCRIPTION:
The aim of this study is to evaluate the tolerability and acceptability of a new plant-based formula for young children. The study population consists of 45 healthy children of ≥12 and <36 months of age

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female children as per the clinical judgement of the Investigator
2. Singleton children
3. Children ≥12 and <36 months of age at screening
4. Children who have been drinking dairy based beverages or plant-based milk replacements (in combination with breastfeeding or not) for at least 3 weeks prior to screening
5. Children are familiar with drinking ≥400 ml/day of dairy based beverages or plant-based milk replacements,
6. Written informed consent from the parent(s) and/or legal guardian(s) (≥ 18 years of age)

Exclusion Criteria:

1. Children with medical conditions requiring a special diet such as fibre-free diet, food allergy, or food intolerances
2. Children with current or previous illnesses/conditions or interventions which could interfere with the study or its outcome parameters (e.g. diarrhoea requiring treatment, constipation requiring treatment, regurgitation requiring treatment, dental/medical procedures which may impact oral feeding), as per the clinical judgment of the Investigator, within 3 weeks prior to screening
3. Use of medication or nutritional/food supplements known to impact GI tolerance (e.g. anti-regurgitation (including any thickening agent), anti-reflux, anti-diarrheal, laxative medication, systemic antibiotic, probiotic supplements) within 3 weeks prior to screening
4. Children who are using diapers
5. Siblings of participating children
6. Participation in any other study involving investigational or marketed products concomitantly or within 3 weeks prior to screening
7. Children of employees and/or family members or relatives of employees of Danone Nutricia Indonesia or of the participating research institute and local community facilities
8. Investigator's uncertainty about the willingness or ability of the parents to comply with the protocol instructions, including daily completion of the diaries by the parents.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Stool characteristics - Stool frequency | Baseline
  Average stool frequency, derived from daily records in the diary
Stool characteristics - Stool frequency | Day 1- 7
  Average stool frequency, derived from daily records in the diary
Stool characteristics - Stool frequency | Day 8- 14
  Average stool frequency, derived from daily records in the diary
Stool characteristics - Stool frequency | Day 15- 21
  Average stool frequency, derived from daily records in the diary
Stool characteristics - Stool consistency | Baseline
  Average stool consistency, derived from daily records in the diary
Stool characteristics - Stool consistency | Day 1-7
  Average stool consistency, derived from daily records in the diary
Stool characteristics - Stool consistency | Day 8-14
  Average stool consistency, derived from daily records in the diary
Stool characteristics - Stool consistency | Day 15-21
  Average stool consistency, derived from daily records in the diary
Stool characteristics - Occurrence of frequent watery stools | Baseline
  Number of watery stools, derived from daily records in the diary
Stool characteristics - Occurrence of frequent watery stools | Day 1-7
  Number of watery stools, derived from daily records in the diary
Stool characteristics - Occurrence of frequent watery stools | Day 8-14
  Number of watery stools, derived from daily records in the diary
Stool characteristics - Occurrence of frequent watery stools | Day 15-21
  Number of watery stools, derived from daily records in the diary
Stool characteristics - Occurrence of hard stools | Baseline
  Number of hard stools, derived from daily records in the diary
Stool characteristics - Occurrence of hard stools | Day 1-7
  Number of hard stools, derived from daily records in the diary
Stool characteristics - Occurrence of hard stools | Day 8-14
  Number of hard stools, derived from daily records in the diary
Stool characteristics - Occurrence of hard stools | Day 15-21
  Number of hard stools, derived from daily records in the diary
Gastrointestinal symptoms | Baseline
  Occurrence of vomiting [present/absent], derived from records in the diary
Gastrointestinal symptoms | Day 1-7
  Occurrence of vomiting [present/absent], derived from records in the diary
Gastrointestinal symptoms | Day 8-14
  Occurrence of vomiting [present/absent], derived from records in the diary
Gastrointestinal symptoms | Day 15-21
  Occurrence of vomiting [present/absent], derived from records in the diary
Flatulence | Baseline
  Occurrence of flatulence [present/absent], derived from records in the diary
Flatulence | Day 1-7
  Occurrence of flatulence [present/absent], derived from records in the diary
Flatulence | Day 8-14
  Occurrence of flatulence [present/absent], derived from records in the diary
Flatulence | Day 15-21
  Occurrence of flatulence [present/absent], derived from records in the diary
Proportion of parents [number / percentage] consulting a health care professional related to medical events linked to gastrointestinal tolerance | Baseline
  Occurrence of parents consulting a health care professional related to medical events linked to gastrointestinal tolerance, derived from records in the diary
Proportion of parents [number / percentage] consulting a health care professional related to medical events linked to gastrointestinal tolerance | Day 1-7
  Occurrence of parents consulting a health care professional related to medical events linked to gastrointestinal tolerance, derived from records in the diary
Proportion of parents [number / percentage] consulting a health care professional related to medical events linked to gastrointestinal tolerance | Day 8-14
  Occurrence of parents consulting a health care professional related to medical events linked to gastrointestinal tolerance, derived from records in the diary
Proportion of parents [number / percentage] consulting a health care professional related to medical events linked to gastrointestinal tolerance | Day 15-21
  Occurrence of parents consulting a health care professional related to medical events linked to gastrointestinal tolerance, derived from records in the diary
Parents' observation and perception of child's wellbeing and stools | Baseline
  Scored as per five-point Danone developed questionnaire ( 1= low satisfaction 5 = high satisfaction) for each of the questions to parents.
Parents' observation and perception of child's wellbeing and stools | Day 1-7
  Scored as per five-point Danone developed questionnaire ( 1= low satisfaction 5 = high satisfaction) for each of the questions to parents.
Parents' observation and perception of child's wellbeing and stools | Day 8-14
  Scored as per five-point Danone developed questionnaire ( 1= low satisfaction 5 = high satisfaction) for each of the questions to parents.
Parents' observation and perception of child's wellbeing and stools | Day 15-21
  Scored as per five-point Likert scale for each of the questions to parents.
Product acceptability | Baseline
  Scored as per five-point Danone developed questionnaire ( 1= low satisfaction 5 = high satisfaction) for each of the questions to parents.
Product acceptability | Day 1-7
  Scored as per five-point Danone developed questionnaire ( 1= low satisfaction 5 = high satisfaction) for each of the questions to parents..
Product acceptability | Day 8-14
  Scored as per five-point Danone developed questionnaire ( 1= low satisfaction 5 = high satisfaction) for each of the questions to parents.
Product acceptability | Day 15-21
  Scored as per five-point Danone developed questionnaire ( 1= low satisfaction 5 = high satisfaction) for each of the questions to parents.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Gadjah Mada, Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No